CLINICAL TRIAL: NCT03358498
Title: Quality of Life and Treatment Satisfaction in β-Thalassemia Patients Receiving Deferasirox
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania, Principal Investigator, Assiut University
Other Study IDs: QOLATSIBTPRD
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: β-thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- β-thalassemia group: SICT It is a questionnaire to assess patient satisfaction with ICT regimens. It comprises 19 items assessing four domains: perceived effectiveness of ICT (PE), burden of ICT (BD), acceptance of ICT (AC), and side effects of ICT (SE). Patients rate all items on scale from 1 "very dissatisfied" to 5 "very satisfied".
  Lab methods :
  1. full history and thorough clinical evaluation.
  2. . Complete blood count. .3- Serum ferritin .
  4-Renal function tests. 5-liver function tests.
  Interventions: Other: The Medical Outcomes Short-Form 36-Item Health Survey (SF-36v2) It

INTERVENTIONS:
Other: The Medical Outcomes Short-Form 36-Item Health Survey (SF-36v2) It — SF-36v2 is questionnaire comprising 36items measuring eight dimensions of general HRQOL: physical functioning 10 items, physical health problems 4 items, bodily pain 2 items, general health perceptions 5 items, vitality 4 items, social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health 5 items.
  .
  Other Names: Satisfaction with ICT Questionnaire (SICT) Complete blood count. - Serum ferritin . -Renal function tests. -liver function tests.

SUMMARY:
Regular blood transfusions are essential for the management of haematological conditions such as β-thalassemia major. As a result, however, patients with these conditions are susceptible to the development of transfusion-dependent iron overload (hemosiderosis or secondary iron overload

DETAILED DESCRIPTION:
In the absence of a naturally occurring physiological mechanism for the removal of excess iron in the body, life-long treatment and adherence to iron chelation therapy (ICT) are necessary to prevent the morbidity and mortality that may result if excess iron is allowed to .

Deferasirox (DFO),is the oldest available form of ICT used by patients with transfusion-dependent disorders. Improvements in ICT administration convenience and tolerability are expected to improve patient's satisfaction with ICT and Health Related Quality of Life (HRQOL), thus promoting adherence to ICT regimens and potentially reducing iron overload-related morbidity/mortality and associated healthcare costs

ELIGIBILITY:
Inclusion Criteria:

1 - Age more than 16 years 2-transfusion related iron over load (serum ferritin more than 1000 ng/ml) 3-patients on oral iron chelation (deferasirox ) for one year or more

Exclusion

1. primary haemochromatosis
2. thalassemia minor patients
3. preseance of systemic disease that prevent patient from treatment ,

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Seventy five thalassemic patients will be included in the study from haematology unit in internal medicine department in Assiut University Hospital.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
The Medical Outcomes Short-Form 36-Item Health Survey (SF-36v2) | Baseline
  - The Medical Outcomes Short-Form 36-Item Health Survey (SF-36v2) It is a self-administered questionnaire comprising 36-items measuring eight dimensions of general HRQOL: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). In addition to scores for individual dimensions, two summary scores assessing physical and mental dimensions of health and well-being can also be calculated: Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Delea TE, Edelsberg J, Sofrygin O, Thomas SK, Baladi JF, Phatak PD, Coates TD. Consequences and costs of noncompliance with iron chelation therapy in patients with transfusion-dependent thalassemia: a literature review. Transfusion. 2007 Oct;47(10):1919-29. doi: 10.1111/j.1537-2995.2007.01416.x. PMID 17880620
- [Background] Bollig C, Schell LK, Rucker G, Allert R, Motschall E, Niemeyer CM, Bassler D, Meerpohl JJ. Deferasirox for managing iron overload in people with thalassaemia. Cochrane Database Syst Rev. 2017 Aug 15;8(8):CD007476. doi: 10.1002/14651858.CD007476.pub3. PMID 28809446
- [Background] Payne KA, Desrosiers MP, Caro JJ, Baladi JF, Lordan N, Proskorovsky I, Ishak K, Rofail D. Clinical and economic burden of infused iron chelation therapy in the United States. Transfusion. 2007 Oct;47(10):1820-9. doi: 10.1111/j.1537-2995.2007.01398.x. PMID 17880607
- [Background] Payne KA, Rofail D, Baladi JF, Viala M, Abetz L, Desrosiers MP, Lordan N, Ishak K, Proskorovsky I. Iron chelation therapy: clinical effectiveness, economic burden and quality of life in patients with iron overload. Adv Ther. 2008 Aug;25(8):725-42. doi: 10.1007/s12325-008-0085-z. PMID 18704280
- [Background] Fisher SA, Brunskill SJ, Doree C, Gooding S, Chowdhury O, Roberts DJ. Desferrioxamine mesylate for managing transfusional iron overload in people with transfusion-dependent thalassaemia. Cochrane Database Syst Rev. 2013 Aug 21;2013(8):CD004450. doi: 10.1002/14651858.CD004450.pub3. PMID 23963793